CLINICAL TRIAL: NCT00592358
Title: Open-Label Study of Invega for the Treatment of Mania in Children and Adolescents Ages 6-17 With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Invega (Paliperidone) for the Treatment of Mania in Children and Adolescents Ages 6-17 With Bipolar Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Associate Professor of Psychiatry at Harvard Medical School and at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-P-001525
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Pediatric Bipolar Disorder
Keywords: bipolar disorder; children; adolescents; Invega
MeSH Terms: conditions — Bipolar Disorder | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: paliperidone

INTERVENTIONS:
Drug: paliperidone — tablet, 3mgQAM - 6mgQAM, taken daily for 8 weeks
  Other Names: Invega

SUMMARY:
This will be an 8-week open-label trial, using daily doses of paliperidone (Invega) in the treatment of children and adolescents who meet DSM-IV criteria of Bipolar I, Bipolar II, or Bipolar Spectrum Disorder. Specific hypotheses are as follows:

Hypothesis 1: Bipolar Disorder symptomatology in children and adolescents with DSM-IV Bipolar I, Bipolar II, or Bipolar Spectrum Disorder will be responsive to Invega treatment.

Hypothesis 2: Invega -associated improvement in bipolar disorder symptomatology in children and adolescents will translate into improved functional capacities (neuropsychological, social, and occupational), as well as an increased quality of life throughout treatment.

Hypothesis 2: Invega treatment will be safe and well tolerated as reflected by a low drop out rate and absence of major side effects.

DETAILED DESCRIPTION:
Invega (paliperidone), a second generation antipsychotic (SGA), is a psychotropic agent belonging to the chemical class of benzisoxazole derivatives. Invega is approved by the FDA for the treatment of schizophrenia in adults. Initial data suggest a promising role for Invega in the treatment of bipolar disorder with minimal adverse events of weight gain. We propose to study the safety and efficacy of Invega therapy in children and adolescents with Bipolar I, Bipolar II, and Bipolar Spectrum Disorder. The study results will be used to generate hypotheses for a larger, randomized, controlled clinical trial with explicit hypotheses and sufficient statistical power.

The proposed study includes 1) use of a 8-week design to document the response rate, 2) assessment of the impact of Invega on functional capacities (quality of life, psychosocial function) and cognition, and 3) careful assessment of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients 6-17 years of age (inclusive).
2. Subjects with the diagnosis of Bipolar or Bipolar Spectrum Disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview. Bipolar Spectrum Disorder (or sub- threshold bipolar disorder) is operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but display fewer elements in Criteria B (only require 2 items for elation category and 3 for irritability).
3. Subjects must score ≥ 20 on the YMRS.
4. Subjects and their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
5. Subjects and their legal representative must be considered reliable reporters.
6. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document (if ≥ 7 years old).
7. Subject must be able to participate in mandatory blood draws.
8. Subject must be able to swallow pills.
9. Subjects with comorbid Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), Obsessive-Compulsive Disorder (OCD), Pervasive Developmental Disorder (PDD), anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of the exclusionary criteria.
10. For concomitant therapy used to treat ADHD, subjects must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the ADHD therapy will not change throughout the duration of the study.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Uncorrected hypothyroidism or hyperthyroidism.
4. Non-febrile seizures without a clear and resolved etiology.
5. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months.
6. Judged clinically to be at serious suicidal risk.
7. Any other concomitant medication with primary central nervous system activity other than specified in the Concomitant Medication portion of the protocol.
8. Current diagnosis of schizophrenia.
9. Mental retardation (IQ < 75).
10. Pregnant or nursing females.
11. Known hypersensitivity to Invega® or similar formulations (paliperidone, risperidone).
12. A non-responder or history of intolerance to Invega®, after treatment at adequate doses as determined by the clinician.
13. Severe allergies or multiple adverse drug reactions.
14. Subjects with a hematological disorder.
15. Subjects with diabetes.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Open label treatment with Invega (Paliperidone) once daily, with dosage of 3mg per day, titrated in 3mg increments to a maximum of 6mg per day based on subject age, weight and tolerance.
Period: Overall Study
Arm/Group | Paliperidone
Started | 17
Completed | 11
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2
Not completed — Inability to swallow pills | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.88 (2.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms Measured by Young Mania Rating Scale (YMRS)
Description: The YMRS is an 11-item instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. Four items are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven itemsare graded on a 0 to 4 scale. The maximum possible total score is 60 (worse outcome, severe symptoms), and the minimum possible total score is 0 (no symptoms).
Time Frame: Baseline and 8 weeks (or final study visit, if subjects completed the study before 8 weeks)
Population: Participants exposed to study medication for a minimum of three weeks were included in analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Paliperidone: Open-label treatment with Paliperidone.
Arm/Group | Paliperidone
Number analyzed (Participants) | 15
units on a scale
  Baseline | 32.8 (6.1)
  Endpoint | 14.1 (11.2)

2. Secondary Outcome: Change in Symptoms Measured by DSM-IV Mania Symptoms Checklist
Description: A 13-item clinician-rated symptom checklist developed by Massachusetts General Hospital to measure symptoms of mania. Each item is given a rating for frequency (1=less than 4 days, 2=greater than or equal to 4 days, 3=daily) and intensity (1=mild, 2=moderate, 3=severe), which are combined to yield a composite severity score ranging from 0 (least severe) to 3 (most severe). The composite severity scores from all 13 items are summed to yield a total measure score, with a minimum score of 0 (least severe) and a maximum score of 39 (most severe).
Time Frame: Baseline and 8 weeks (or final study visit, if subjects completed the study before 8 weeks)
Population: All participants for whom the mania checklist was available at both baseline and endpoint (8-weeks) were included in analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone
Number analyzed (Participants) | 8
units on a scale
  Baseline | 18.5 (5.6)
  Endpoint | 10.9 (6.3)

ADVERSE EVENTS:
Arm/Group | Paliperidone
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone (N=15)
Plaque-like skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Superficial scratches on arm (Skin and subcutaneous tissue disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1)
Mild extrapyrimidal symptoms (General disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2)
Eye twitching (Eye disorders) | 1 (2)
Flu like symptoms (General disorders) | 3 (3)
Headache (General disorders) | 3 (7)
Increased appetite (Metabolism and nutrition disorders) | 6 (15)
insomnia (General disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 1 (3)
Heart palpitation (Cardiac disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (6)
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Strep throat (General disorders) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Worsening of anxiety and depressive symptoms (Psychiatric disorders) | 1 (1)
Low appetite (Metabolism and nutrition disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes